CLINICAL TRIAL: NCT05028374
Title: Phase II Trial Evaluating the Efficacy of Moderna COVID-19 Vaccine Booster Dosing in Patients With Hematologic Malignancies Who Did Not Have an Adequate Response to Prior Vaccination
Brief Title: COVID-19 VAX Booster Dosing in Patients With Hematologic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Jeffrey Zonder, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-036
Record Dates: First submitted 2021-08-23; First posted 2021-08-31 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-11

CONDITIONS: Multiple Myeloma; AL Amyloidosis; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Multiple Myeloma; Immunoglobulin Light-chain Amyloidosis; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- A single "booster" dose of the Moderna mRNA COVID-19 vaccine administered intramuscularly (Other): The dose of Moderna mRNA vaccine to be administered is the same for all patients in all enrollment cohorts: 0.5 mL administered intramuscularly as a single dose, according to the manufacturer's package insert.
  Interventions: Drug: A single "booster" dose of the Moderna mRNA COVID-19 vaccine

INTERVENTIONS:
Drug: A single "booster" dose of the Moderna mRNA COVID-19 vaccine — All participants will receive a single dose of the Moderna mRNA COVID-19 vaccine administered intramuscularly. This is an open label, non-randomized trial.
  Other Names: Covid 19 booster dose

SUMMARY:
To determine whether protective antibody levels increase after booster dosing with the Moderna COVID-19 vaccine in patients diagnosed with Hematologic Malignancies who have low antibody levels after a prior first vaccination with any of the SARS-CoV2 vaccines that were authorized for use in the USA. Researchers will also assess whether the booster dosing with the Moderna COVID-19 vaccine is safe in patients with multiple myeloma, amyloidosis, or other blood cancers.

DETAILED DESCRIPTION:
The specific hypothesis being tested is that it may be possible to induce a protective humoral immune response with a booster dose of the Moderna COVID-19 vaccine in patients with hematologic malignancies who did not have an adequate response to first vaccination with any of the available COVID-19 vaccines. To test this hypothesis, t a Phase II singlestage trial in which patients with a negative or weak positive anti-SARS-CoV2 IgG antibody test (defined as <1.00 S/CO and 1.00-1.99 S/CO, respectively) will receive a single standard dose of the Moderna COVID-19 vaccine intramuscularly, and then have anti-SARS-CoV2 IgG antibody levels checked 28 days (+/-3 days) later.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 years of age or older
4. Previously diagnosed with MM/AL amyloidosis (Cohorts 1 or 3) or other hematologic malignancy (Cohorts 2 or 3).
5. Previously received any one of the available COVID-19 vaccines (between 4 and 36 weeks prior to enrollment)
6. Anti-SARS-CoV2 IgG antibody titer of results less than 1.0 units (Cohorts 1 and 2), or 1.0-1.99 units (Cohort 3). Antibody titers will be measured within 14 days of enrollment.
7. If currently receiving potentially immunosuppressive anti-neoplastic therapy for their underlying hematologic condition, a two-week interruption in therapy before and after the booster dose of vaccine is ENCOURAGED BUT NOT REQUIRED (physician discretion).-

Exclusion Criteria:

1. Daily corticosteroids at a dose equivalent to Prednisone 20 mg/day or greater during the period two weeks before enrollment to the trial. Intermittent steroid dosing at or above this level is permitted (i.e., weekly dexamethasone dosing as part of myeloma therapy)
2. History of previous severe reaction to any available COVID-19 vaccine (defined as any Grade 3 or higher reaction)
3. Febrile illness within 3 days of booster dosing.
4. Documented SARS-CoV2 infection within 2 weeks of enrollment.
5. Less than 3 months post-autologous or allogeneic stem cell transplant (NOTE: transplant between initial standard vaccine administration and enrollment is NOT otherwise grounds for exclusion from participation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Zonder, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Multiple myeloma and amyloidosis patients who did not develop an anti-spike antibody titer of >1 S/CO after prior COVID-19 vaccination.
- Cohort 2: Patients with other hematologic malignancies who did not develop an anti-spike antibody titer of >1 S/CO after prior COVID-19 vaccination.
- Cohort 3: Patients with multiple myeloma, amyloidosis, or other hematologic malignancy who had a "weak positive" response to prior COVID-19 vaccine, defined as an anti-spike antibody titer of 1-2 S/CO.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 52 | 51 | 16
Completed | 52 | 50 | 16
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 52 | 51 | 16 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 18 | 10 | 43
  >=65 years | 37 | 33 | 6 | 76
Age, Continuous [Median (Full Range); unit: years] | 68 [45 to 94] | 68 [35 to 92] | 63.5 [32 to 82] | 68 [32 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 18 | 6 | 49
  Male | 27 | 33 | 10 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 7 | 2 | 12
  White | 49 | 43 | 12 | 104
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Observed Response Rate of Anti-SARS-CoV2 Antibody Seroconversion.
Description: Anti-SARS-CoV2 IgG antibody seroconversion from negative to positive.
Time Frame: 28 days (+/- 3 days) following a booster dose of the Moderna mRNA COVID-19 vaccine
Population: Participants who received a single dose of the Moderna mRNA COVID-19 vaccine administered intramuscularly.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 52 | 50 | 16
Participants | 29 | 28 | 0

2. Secondary Outcome: Observed Rate of STRONG POSITIVE Anti-SARS-CoV2 Antibody Response
Description: A STRONG POSITIVE response is defined in this trial as an anti-SARS-CoV2 IgG antibody titer of at least 2 S/CO 28 days (+/- 3 days) following vaccine administration
Time Frame: measured 28 days (+/- 3 days) following a booster dose of the Moderna COVID-19 vaccine.
Population: Participants who received a single dose of the Moderna mRNA COVID-19 vaccine administered intramuscularly.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 52 | 50 | 16
Participants | 27 | 23 | 15

ADVERSE EVENTS:
Time Frame: Daily phone calls or video chats for 1 week following vaccine administration, and then weekly after that until 4 weeks after vaccination.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 6/52 | 4/50 | 2/16
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/50 | 1/16
Other Adverse Events (participants affected / at risk) | 48/52 | 47/50 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=52) | Cohort 2 (N=50) | Cohort 3 (N=16)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=52) | Cohort 2 (N=50) | Cohort 3 (N=16)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Cardiac disorders - Other (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (7) | 3 (6) | 2 (2)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 4 (4) | 1 (1) | 1 (1)
Edema limbs (General disorders) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 12 (13) | 20 (21) | 8 (8)
Fever (General disorders) | 3 (3) | 3 (3) | 4 (5)
Injection site reaction (General disorders) | 36 (37) | 40 (43) | 16 (16)
Irritability (General disorders) | 1 (1) | 0 (0) | 0 (0)
Localized edema (General disorders) | 2 (2) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Investigations - Other (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (10) | 12 (13) | 8 (8)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 6 (6) | 7 (8) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/74/NCT05028374/Prot_SAP_000.pdf